CLINICAL TRIAL: NCT04074486
Title: Evaluation and Validation of a Multimodal Brain Function Biomarker With NPC
Acronym: BSC-CI-NPC
Status: Completed | Type: Observational
Sponsor: BrainScope Company, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 55/60
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Brain Injuries; Concussion, Mild; Concussion, Brain; Near Point Convergence; Concussion, Intermediate
Keywords: Concussion; Mild Traumatic Brain Injury; Automated/Electronic Near Point Convergence
MeSH Terms: conditions — Brain Injuries; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Injured and Matched Control Subjects: Head Injured subjects are defined as those who sustained a closed head injury and meet specified protocol inclusion/exclusion criteria. Matched Control subjects are enrolled based on matching criteria (for e.g. age, gender, and same population i.e. sports vs non-sports) to the head injured subjects. For all head injured and matched control group subjects, the full battery of tests will be performed. The injured pool will begin test procedures when a subject sustains a concussion injury. The matched control pool will follow the same time point/date interval as their matched injured subject. The matched control will be assigned by site to an injured subject and matched by age, gender, and sport (if applicable) or from the same population (if non-sport).
  Interventions: Device: BrainScope Ahead 300iP-O; Diagnostic Test: SCAT5; Diagnostic Test: Near Point Convergence
- Healthy Volunteer Subjects: Healthy Volunteer subjects are defined as those who are normal subjects i.e. not head-injured meeting specified protocol inclusion/exclusion criteria.This group of subjects are recruited only for the purpose of collecting data for norming the electronic near point convergence measurement (eNPC). These subjects will only perform a limited battery of BrainScope tests at a single visit and will include data collection regarding their demographics, concussion history, signs and symptoms, sports information, etc. These subjects will not undergo EEG or neurocognitive assessment.
  Interventions: Device: BrainScope Ahead 300iP-O; Diagnostic Test: SCAT5; Diagnostic Test: Near Point Convergence
- Non-Concussed Head Injured Subjects: A secondary group of non-concussed head-injured controls shall be also recruited who were observed to have a head impact/injury but were not restricted from play within the same game or deemed non-concussed following on-field/sideline evaluation by the standard of care at each site. They will perform the entire BrainScope battery of tests within 5 days after the incident and defined as Day 0 and a follow-up assessment at 15 Days following Day0
  Interventions: Device: BrainScope Ahead 300iP-O; Diagnostic Test: SCAT5; Diagnostic Test: Near Point Convergence

INTERVENTIONS:
Device: BrainScope Ahead 300iP-O — BrainScope study battery consists of four components: recording of brain electrical activity (EEG); three neurocognitive performance tests; an electronic Near Point Convergence measurement assessment and clinical symptom assessments.
Diagnostic Test: SCAT5 — Sports Concussion Assessment Tool 5
Diagnostic Test: Near Point Convergence — Manual ocular function measurement conducted only if electronic version on device fails

SUMMARY:
This study is designed to collect data which will be used to associate changes in EEG, neurocognitive performance, eNPC and clinical symptoms in concussion subtypes. The study will recruit males and females, 13-50 years old, from Concussion Centers/Programs, Sports Venues and Emergency Departments (ED) across the country, over an 18-month period (Phase 2, 12 months for Algorithm Development and Norming, and Phase 3, 6 months for Validation).

DETAILED DESCRIPTION:
Phase 1 of this project (USAMRDC W81XWH-18-C-0157) was focused on building the automated/electronic NPC capability (eNPC). This protocol is for Phase 2, in which the CI multimodal brain function biomarker will be extended (Algorithm Development) with the inclusion of an automated ocular function measurement (AOFM), to expand the capability in the characterization of concussion. The study will also expand the range of applicability of the CI to ages 13-50 years old. Phase 2 will also include norming of eNPC across the age range. Phase 3 of the project will validate the algorithms developed in Phase 2, using the same protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥13 and <51 years old at time of enrollment;
* No prior history of concussion or TBI in the last 6 months.

For head injured subjects

* Having sustained a traumatic closed head injury within 120 hours (5 days from time of injury at time of BrainScope assessment);
* GCS 13-15 at time of BrainScope assessment.

For non-concussed head-injured controls

* Having sustained a traumatic closed head injury but returned to play or deemed non-concussed following sideline (on-field) evaluation within the same game and enrolled in the study within 120 hours (5 days) from said incident.
* GCS 13-15 at time of BrainScope assessment.

For matched controls and healthy volunteers

• GCS 15 at time of BrainScope assessment.

Exclusion Criteria:

* Enrolled in any previous BrainScope clinical study;
* Current CNS active prescription medications taken daily, except for medication being taken for the treatment of Attention Deficit Disorders (ADD/ADHD); medication for smoking cessation; or medications for anxiety taken PRN (as needed);
* Forehead, scalp or skull abnormalities that prevents headset application for EEG data collection in injured/matched controls;
* History of brain tumor, brain surgery or known neurological disease including, Parkinson's, MS, Alzheimer's, dementia, epilepsy;
* History of TIA or Stroke within the last year;
* Pregnant women;
* Subjects who do not speak English (non-English speaking parents are allowed to consent so long as translation of the consent form in their native language is available);
* Acute intoxication ;
* Evidence of illicit drug abuse in the last year;
* Active fever defined as greater than 100ºF or 37.78ºC at time of BrainScope assessment;
* Subjects currently receiving dialysis or have end-stage renal disease;
* Subjects requiring advanced airway management (i.e. mechanical ventilation);
* Prisoners.

For head injured subjects

* Loss of consciousness ≥ 20 minutes related to the concussion injury;
* Evidence of abnormality visible on Computerized Tomography (CT) of the head related to the traumatic event (note: neuroimaging is not required for enrollment);
* For current injury, hospital admission (other than the Observation Unit) ranging more than 24 hours due to either head injury or collateral injuries.

For non-concussed head-injured controls

* Loss of consciousness ≥ 20 minutes related to the head impact;
* Any focal neurological signs including aphasia, apraxia, diplopia, facial droop, dysarthria/slurred speech;
* Any score >3 on a 7-point Likert scale (0=none, 6=severe) for the following symptoms at the time of BrainScope assessment (compared to how the subject normally feels): headache, dizziness, balance problems, neck pain, feeling slowed down;

For matched controls and healthy volunteers

* Any focal neurological signs including aphasia, apraxia, diplopia, facial droop, dysarthria/slurred speech;
* Hospital admission (other than the Observation Unit) ranging more than 24 hours due to either head injury or collateral injuries in the past 6 months;
* Any score >3 on a 7-point Likert scale (0=none, 6=severe) for the following symptoms at the time of BrainScope assessment (compared to how the subject normally feels): headache, dizziness, balance problems, neck pain, feeling slowed down.

For healthy volunteers

* Legally blind in one or both eyes;
* History of eye surgery in the past year;
* Any known eye disorders including age-related macular degeneration (AMD), glaucoma, lazy eye, diplopia, cataracts, etc.

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Male and female study subjects aged 13-50 from participating sites will be invited to enroll the study.
Sampling Method: Non-Probability Sample
Enrollment: 1318 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the multivariate and multimodal Concussion Index | 18 months for data acquisition
  Sensitivity and specificity of the expanded CI for assessment of the likelihood of concussion in subjects ages 13-50 who sustained a closed head injury.

SECONDARY OUTCOMES:
Efficacy of use | 18 months for data acquisition
  The demonstration of efficacy of use of this biomarker of brain function impairment/concussion to assess readiness to return to normal activity
Identification of concussion subtypes | 18 months for data acquisition
  Validation of subtypes (at time of injury) with different clinical characterizations and outcome (e.g., rapid versus prolonged recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Prichep, Ph.D., Study Director — BrainScope Company, Inc.
Locations (6):
- United States (6):
  - University of Arkansas, Fayetteville, Arkansas
  - University of Connecticut, Storrs, Connecticut
  - University of Miami, Miami, Florida
  - Michigan State University, East Lansing, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - INOVA Health System, Fairfax, Virginia